CLINICAL TRIAL: NCT04693884
Title: The Influence of Cannabis Inhalation During Exercise on Cardiovascular Health and Function: Exploring the Optimal Balance of Cannabinoids and Mode of Administration to Decrease Risk and Maximize Benefits
Brief Title: Cannabis Inhalation: Effects on Cardiovascular Function During Rest and Exercise
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jamie Burr (Other)
Responsible Party: Sponsor-Investigator, Jamie Burr, Associate Professor, University of Guelph
Organization: University of Guelph (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UOG-HPL-CAN (REB# 18-11-013)
Record Dates: First submitted 2020-11-03; First posted 2021-01-05 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Cannabis; Cardiovascular Risk Factor
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High THC, Smoked (Experimental)
  Interventions: Drug: Cannabis
- High THC, Vaporized (Experimental)
  Interventions: Drug: Cannabis
- High CBD, Smoked (Experimental)
  Interventions: Drug: Cannabis
- High CBD, Vaporized (Experimental)
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Cannabis of (~10% THC concentration <1% CBD concentration) will be smoked.
  Other Names: High THC, Smoked
  Arms: High THC, Smoked
Drug: Cannabis — Cannabis of (~10% THC concentration <1% CBD concentration) will be vaporized.
  Other Names: High THC, Vaporized
  Arms: High THC, Vaporized
Drug: Cannabis — Cannabis of (~10% CBD concentration <1% THC concentration) will be smoked.
  Other Names: High CBD, Smoked
  Arms: High CBD, Smoked
Drug: Cannabis — Cannabis of (~10% CBD concentration <1% THC concentration) will be vaporized.
  Other Names: High CBD, Vaporized
  Arms: High CBD, Vaporized

SUMMARY:
This two-phase project seeks to examine the cardiovascular response to consumption of cannabis variants of different cannabinoid composition through different methods (smoking vs. vaporizing), at rest and during aerobic exercise. Multiple measures that have been shown to predict risk factors for chronic-disease and negative health outcomes will be assessed following cannabis consumption at rest or in combination with exercise. These techniques will examine arterial stiffness, vascular function, and cardiac function. In phase I and II, subjects will visit the lab on 6 different occasions; with 1 visit acting as an introductory visit, 1 as an exercise control visit, 2 as resting cannabis visits, and 2 as cannabis + exercise visits. Cannabis used in phase I of this study will consist of approximately 10% THC. On all visits, pulse wave velocity, flow mediated dilation, and echocardiography measures will be performed following cannabis consumption by smoking or vaporizing, and cannabis consumption by smoking or vaporizing followed by 20 minutes of exercise on a cycle ergometer. Phase II of the study will implore a similar design. In favor of altering method of consumption, in all visits cannabis will be consumed by vaporization and will be either a high cannabidiol (CBD: (~10%)) and low delta-9-tetrahydrocannabinol (THC: (<1%)), or a high THC (~10%) and low CBD (<1%) variant.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 19-45yr
4. In good general health as evidenced by medical history and free of chronic disease
5. Must be experienced with cannabis use. This requires recreational cannabis use of a minimum of once per week in the past 30 days as confirmed by urine test
6. Experience consuming cannabis recreationally by vaping dried cannabis

Exclusion Criteria:

1. Deemed unfit to exercise by the PARQ+.
2. Current or past diagnoses of substance abuse disorder
3. Failure of recreational substance urine screening test
4. Current, past, or strong family history of psychosis, or has previously experienced a cannabis-related psychotic episode
5. Current or past diagnoses of cannabis use disorder
6. Current or past diagnoses of any mood or anxiety disorder
7. Identified ECG abnormalities
8. Systolic blood pressure exceeding 160mmHg
9. Diastolic blood pressure exceeding 90mmHg
10. Resting heart rate exceeding 100bpm, or lower than 40bpm
11. Diagnosed with respiratory disease
12. Diagnosed with cardiovascular disease
13. Diagnosed with liver disease
14. Diagnosed with kidney disease
15. Is Pregnant or planning to be pregnant
16. Currently taking prescription medication (excluding contraceptive medication)
17. Is a cigarette smoker

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Change in Aortic Stiffness From Baseline Following Cannabis Consumption | Baseline, Post-Intervention (<2 Hours)
  Assessed via carotid-femoral pulse wave velocity (PWV)
Change in Brachial Artery Vascular Function From Baseline Following Cannabis Consumption | Baseline, Post-Intervention (<2 Hours)
  Assessed via brachial artery flow mediated dilation (FMD)
Change in Sympathetic Nervous System Activity From Baseline Following Cannabis Consumption | Baseline, Post-Intervention (<2 Hours)
  Assessed via microneurographic recordings of the peroneal nerve
Change in Cardiac Function From Baseline Following Cannabis Consumption | Baseline, Post-Intervention (<2 Hours)
  Measured by echocardiography

SECONDARY OUTCOMES:
Exercise Capacity | Baseline, Post-Intervention (<2 Hours)
  Assessed by maximal average power attainable during 20 minutes of continuous cycling exercise
Heart Rate | Baseline, Post-Intervention (<2 Hours)
  Measured at rest and during exercise
Systolic Blood Pressure | Baseline, Post-Intervention (<2 Hours)
  Measured at rest and during exercise
Diastolic Blood Pressure | Baseline, Post-Intervention (<2 Hours)
  Measured at rest and during exercise
Perceived Exertion | Baseline, Post-Intervention (<2 Hours)
  Measured during exercise
Oxygen Consumption | Baseline, Post-Intervention (<2 Hours)
  Measure of metabolic activity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cheung CP, Coates AM, Baker RE, Burr JF. Acute Effects of Cannabis Inhalation on Arterial Stiffness, Vascular Endothelial Function, and Cardiac Function. J Am Heart Assoc. 2024 Dec 3;13(23):e037731. doi: 10.1161/JAHA.124.037731. Epub 2024 Nov 22. PMID 39575727
- [Derived] Cheung CP, Nardone M, Lee JB, Baker RE, Millar PJ, Burr JF. Cannabis Inhalation Acutely Reduces Muscle Sympathetic Nerve Activity in Humans. Circulation. 2022 Dec 20;146(25):1972-1974. doi: 10.1161/CIRCULATIONAHA.122.062564. Epub 2022 Oct 31. No abstract available. PMID 36314198

DOCUMENTS (2):
  • Study Protocol (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT04693884/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT04693884/SAP_001.pdf